CLINICAL TRIAL: NCT01118247
Title: Primary Uncemented Total Hip Prosthesis With Pure Ti With and Without HA, and Alumina-on-alumina Articulation
Brief Title: Primary Uncemented Partly Ti-coated Total Hip Prosthesis With and Without HA, and Alumina-on-alumina Articulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-REK NORD 44/206; 200602701-8/IAY/400 (Other: North Norwegian Ettic Commitee)
Record Dates: First submitted 2010-04-30; First posted 2010-05-06 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Survival of the Implants With Revision as Endpoint; Clinical Performance With HHS; Patients Satisfaction With the Hip Implant
Keywords: Uncemented THA; alumina-on-alumina; survival; HHS; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pure Ti (Experimental): Cup and stem partly coated with pure titanium
  Interventions: Procedure: Uncemented primary total hip arthroplasty
- pure Ti and HA (Active Comparator): Cup and stem partly coated with pure titanium, and fully coated with HA.
  Interventions: Procedure: Uncemented primary total hip arthroplasty

INTERVENTIONS:
Procedure: Uncemented primary total hip arthroplasty — Total hip prosthesis partly coated with pure Ti with and without HA are compared in a RCT.
  Other Names: Cup: Igloo, Biotechni, Fr; Stem: Filler, Biotechni, Fr; Head, liner: Biotechni, Fr, Morgan, GB

SUMMARY:
Both HA coated and certain uncoated femoral stems have good results in general. On the cup side the results are more variable, either with or without HA. HA may delaminate from the prosthesis, damage the articulation, witch may lead to osteolysis and aseptic loosening.

The investigators are investigating whether a well working uncemented hip prosthesis design with HA coating, will perform without HA in the long run, when the investigators use pure Ti macrostructure and alumina on alumina articulation.

Hypothesis: The bone ingrowth will be equal when the surface has almost equal roughness in Ti and HA version. This means that HA on Ti is not necessary with a well functioning prosthesis design.

0-hypothesis:The two prosthesis perform equal in survival, clinically (HHS),radiographic and in patient satisfaction at 2, 5, 10, 15 and 20 years.

DETAILED DESCRIPTION:
Investigate survival of the implants and possible biological consequences. Clinical outcome with Harris Hip Score. Radiographic outcome with a modified protocol after JRC, JBJS 1990. Patient satisfaction with the hip prosthesis (five categories).

Grit blasted TiAL6V4 + pure Ti versus grit blasted TiAL6V4 + pure Ti +HA, with almost the same roughness. Screw cup, double tapered stem, partly double coated cup, proximally double coated stem.

Prospective RCT. Multicenter ( Three hospitals). Selected surgeons. Non-inferiority-design.

At present 569 hips (391 patients, 178 bilateral) are randomized into the study. Inclusion of patients into the study stopped in January 2013.

548 hips have completed follow ups at an average of 2 years, 301 hips have completed follow ups at an average of 5 years and 60 hips at 8-10 years.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary osteoarthrosis.
* Both gender, less than seventy years.
* Patients operated for FCF and patients with previous osteotomies are included.

Exclusion Criteria:

* Treatment with Prednisolon.
* Osteomyelitis.
* Serious infections illnesses.
* Cancer or metastasis.
* Rheumatoid arthritis.
* Osteonecrosis after use of alcohol or medicaments.
* Kidney illnesses.
* Metabolic bone diseases.
* Earlier hip arthrodesis.
* Allergic reactions on implants.
* Patients who do not cooperate on rehabilitation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2004-04; Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Survival with revision as endpoint. | 5-20 years

SECONDARY OUTCOMES:
Clinical outcome with Harris Hip Score. | 10-30 years
Radiographic outcome. | 10-30years
  The radiographic evaluation will be carried out postoperatively, 2, 5, 10, 15 and 20 years after the operations with the same protocol modified after Johnston et al, JBJS Am. 1990;72: page 166. We judge and compare a.p pelvic x-rays calibrated on the computer.
Patient satisfaction with the hip prosthesis. | 10-30 years
  At the consultations we ask the patient if he/she is satisfied with the hip. The patient may answer i 5 categories (dissatisfied, not satisfied, satisfied, very satisfied and very much satisfied). We also have registrations on early and late complications, leg length discrepancy, Trendelenburg lurch etc.

CONTACTS AND LOCATIONS:
Overall Officials: Olav Reikerås, MD, Prof, Study Director — Department of Orthopaedics, Rikshospitalet University Clinic, University of Oslo, N-0027 Oslo, Norway.; Arvid Småbrekke, MD, Principal Investigator — University Hospital of North Norway
Locations (1):
- Ortopaedic Department, University Hospital of North Norway, Tromsø, Norway